CLINICAL TRIAL: NCT00682409
Title: Magnetic Resonance (MR) Imaging in the Post Operative Follow-up of Cholesteatoma in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007-A00743-50; 2007-22
Record Dates: First submitted 2008-05-16; First posted 2008-05-22 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Cholesteatoma
MeSH Terms: conditions — Cholesteatoma | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Analysis of the value of the imaging of distribution and the late sequence to differentiate the cholesteatoma of the fibrosis in the follow-up operating post at the child
  Interventions: Other: MR Imaging

INTERVENTIONS:
Other: MR Imaging — MR imaging in the post operative follow-up of cholesteatoma in children

SUMMARY:
Classical imaging techniques are inaccurate to detect residual cholesteatoma. The aim of our study is to evaluate the value of diffusion-weighted MR imaging and delayed contrast enhanced T1 weighted spin-echo sequences in the detection of residual cholesteatoma in children, in a large serie of surgically verified cases.

DETAILED DESCRIPTION:
Classical imaging techniques are inaccurate to detect residual cholesteatoma. Thin-section CT detects that the postoperative cavity is filled with a soft tissue mass. Classical MR imaging (T2 and T1 weighted spin-echo sequences) can not provide additionnal information about the nature of this filling : cholesteatoma, granulation or fibrous tissue.

ELIGIBILITY:
Inclusion Criteria:

* Female or male child enters 5 and 18 years
* Child having benefited from a surgical operation for cholesteatoma of the average ear acquired or congenital, one-sided or bilateral
* Child for whom an additional operating time is indicated
* Child without contraindication in the MRI
* Child having signed a enlightened assent
* Child among whom the parents or the legal representatives signed a enlightened assent

Exclusion Criteria:

* Child of less than 5 years old and more than 18 years
* Child presenting a chronic renal insufficiency
* Child for whom an additional operating time is not indicated
* Child having a contraindication in the MRI
* Child not having signed the assent or the parents of which did not sign the assent

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2008-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Technical characteristics of the examination MRIs represented by the sensibility and the specificity of the test, with regard to the results stemming from the surgical operation | 24 months

SECONDARY OUTCOMES:
Only a surgical operation will confirm the diagnosis of cholesteatoma doing it again or residual. | 24 months
It is necessary to test the following diagnostic method: the analysis of the morphological sequences in T1 and in T2 will allow to appreciate the existence or not of a filling of the cavity tympanique or the mastoïde and to clarify its localization. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte BOURLIERE NAJEAN, MD, Principal Investigator — Assistance Publique des Hôpitaux de Marseille
Locations (1):
- Hôpital de la Timone- Service de radiologie pédiatrique et d'ORL pédiatrique, Marseille, France